CLINICAL TRIAL: NCT04996927
Title: A Prospective, Single-arm, Observational Clinical Study Based on 18F-FDG PET/CT to Evaluate the True Efficacy and Immune Response of PD-1 Monoclonal Antibody Combined With First-line Chemotherapy in Advanced Non-small Cell Lung Cancer
Brief Title: 18F-FDG PET/CT to Evaluate pD-1 Monoclonal Antibody With First-line Chemotherapy in Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan-0200
Record Dates: First submitted 2021-06-27; First posted 2021-08-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a diagnostic study. Subjects were enrolled from clinical stage IIIB or IV NSCLC patients who received standard first-line chemotherapy combined with PD-1 monoclonal antibody immunotherapy and received 18F-FDG PET/CT imaging before treatment, after 2 courses of treatment, and at the time of disease progression.At the same time, the blood routine, liver and kidney function, inflammatory indexes and other laboratory data of the subjects participating in the study were collected. Based on 18F-FDG PET Ipercist standard and comprehensive laboratory indicators, the subjects were evaluated for tumor biological characteristics prediction and clinical staging, PD-1 immune efficacy monitoring and evaluation, tumor recurrence monitoring and re-staging. At the same time, the systemic immune response and immune-related adverse events during the treatment process were evaluated in order to establish a better evaluation standard and system for the comprehensive evaluation of PD-1 immunotherapy.This study plans to set the sample size as 50 cases.

DETAILED DESCRIPTION:
This is a diagnostic study. Subjects were enrolled from clinical stage IIIB or IV NSCLC patients who received standard first-line chemotherapy combined with PD-1 monoclonal antibody immunotherapy and underwent 18F-FDG PET/CT imaging before treatment, after two lines of treatment and at the time of disease progression, while routine blood counts, liver and kidney function, inflammatory indices and other laboratory data were collected from subjects enrolled in the study. Based on standard 18F-FDG PET Ipercist and comprehensive laboratory indicators, subjects were evaluated for prediction of tumour biological characteristics and clinical staging, monitoring and evaluation of PD-1 immune efficacy, monitoring of tumour recurrence and restaging. At the same time, the systemic immune response and immune-related adverse events during the treatment process were evaluated to establish a better evaluation standard and system for the comprehensive evaluation of PD-1 immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or above), gender unlimited;
* Pathological diagnosis of non-small cell lung cancer stage IIIB or above;
* Agree to carry out the standard first-line chemotherapy combined with immunosuppression established in this study;
* Consent to 18F-FDG PET/CT imaging and related laboratory examination before and during treatment;
* The patients themselves or their legal representatives are aware of this study and can sign the informed consent.

Exclusion Criteria:

* Acute systemic diseases and electrolyte disturbances;
* Pregnant or lactating women;
* The patient or his legal representative is unable or unwilling to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed stage IIIb-IV non-small cell lung cancer (according to the International Association for the Study of Lung Cancer Chest Tumor Staging Manual, Edition 7. IASLC Staging Manual in Thoracic Oncology. The patient's tumor must lack an EGFR-sensitive mutation (i.e. exon 19 deletion, or exon 21 L858R, exon 21 L861Q, exon 18 G719X, or exon 20 S7681 mutation) and ALK rearrangement.Patients must provide a biopsy for PD-L1 testing. The World Health Organization (WHO)/ Eastern Collaborative Oncology Group (ECOG) physical status score was 0 or 1 at the time of enrollment. At least 1 lesion (no previous radiotherapy) whose longest diameter ≥10mm was accurately measured by CT or MRI at baseline. Must have a life expectancy of at least 12 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 18F-FDG PET/CT for diagnosis the true efficacy and immune response of Non-small Cell Lung Cancer | 2 years
  PET/MR results will be compared with histopathological, clinical, laboratory, radiological evidence, and follow-up results.

SECONDARY OUTCOMES:
Change after treatment | 2 years
  For patient after treatment, change of PET scan and clinical/radiological/histopathological indices.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China